CLINICAL TRIAL: NCT00411411
Title: Phase 3, Double Blinded, Placebo Controlled Study of the Effects of 12 Weeks DPP-IV Inhibitor Treatment on Secretion and Action of the Incretin Hormones in Patients With Type 2 Diabetes
Brief Title: Long Term Effects of DPP-IV Inhibitor Treatment in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Kasper Aaboe, Doctor, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1502
Record Dates: First submitted 2006-12-13; First posted 2006-12-14 (Estimated); Results first posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-07

CONDITIONS: Type 2 Diabetes
Keywords: GLP-1; GIP; Incretin hormones; DPP-IV inhibitor; Hyperglycaemic clamp; Meal test
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo treatment, administered as tablets.
  Interventions: Drug: Placebo
- Januvia (Experimental): Active treatment
  Interventions: Drug: Januvia

INTERVENTIONS:
Drug: Januvia — 200 mg t.i.d
  Other Names: Sitagliptin
  Arms: Januvia
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
We wish to evaluate the effect of long term treatment with a DPP-IV inhibitor on the function of the incretin hormones

Hypothesis We hypothesize that that a gradual improvement in metabolic control induced by DPP-IV inhibitor (Januvia®) treatment significantly ameliorates the impaired secretion and potency of GLP-1 and leads to a restoration of the lost action of GIP.

DETAILED DESCRIPTION:
Background The incretin effect, primarily mediated by the peptide hormones GIP and GLP-1, is known to be impaired in patients with type 2 diabetes, and characterised by reduced GLP-1 secretion and potency and a lack of responsiveness to the insulinotropic effect of GIP. The cause of this defect remains unknown, but exogenous administration of GLP-1 has shown promising results in attempts to restore the incretin effect. Due to rapid degradation of both incretin hormones by the enzyme dipeptidyl-peptidase IV (DPP-IV), treatment strategies now focus on GLP-1 analogues and prevention of hormone degradation through DPP-IV inhibition.

Hypothesis We hypothesize that that a gradual improvement in metabolic control induced by DPP-IV inhibitor (Januvia®) treatment significantly ameliorates the impaired secretion and potency of GLP-1 and leads to a restoration of the lost action of GIP.

Objective To assess the effect of three months treatment with Januvia®, administered as tablets once daily, on metabolic control in metformin treated patients with type 2 diabetes, measured as increases in incretin hormones and insulin secretion.

Efficacy end points Primary efficacy end point in trial part one is the relative increase in meal-induced total GLP-1 secretion after one and twelve weeks of Januvia® treatment.

Primary efficacy end point in part two is restoration of the insulinotropic effect of GIP, measured as the relative increase in GIP induced amplification of the late phase insulin secretion (AUC) response to glucose after 12 weeks of Januvia® treatment.

Secondary objectives are examination of GLP-2, somatostatin, glucagon, peptide-YY and two glycaemic control parameters (HbA1c and fasting plasma glucose)

Design This is a single centre, randomized, double blinded, placebo controlled trial. The trial consists of two parts, each consisting of three months of inhibitor treatment. In each part, 24 patients, recruited from the Diabetes Outpatient Clinic of Gentofte University Hospital, will be randomized to a treatment supplement of either Januvia® or placebo.

Procedures During the trial, patients will be tested with well established procedures. In part one, patients will undergo a standardized meal test and two β-cell secretory capacity tests. In part two, patients will undergo standardized hyperglycaemic GIP, GLP-1 and saline clamps.

Safety The trial has a short time span of only three months. With more than ten visits during this time and regular blood sampling, the patients are well monitored.

ELIGIBILITY:
Inclusion criteria

* Type 2 diabetes diagnosed according to and in accordance with the WHO criteria
* Metformin treatment of ≥ 1 gram
* 7,5 % ≤ HbA1c ≤ 10%
* Age > 18
* BMI ≥ 25 kg/m2
* Informed consent
* Contraception, if appropriate

Exclusion criteria

* Proliferating retinopathy
* Uremia, end stage renal disease, diabetic nephropathy or any other cause of impaired renal function with s-creatinine > 130 µM and/or albuminuria (>300 mg/day)
* Liver disease with ALAT and/or ASAT > 2 x normal value
* Complicated coronary artery disease, NYHA group III and IV
* Positive screening for islet cell auto antibodies and/or GAD-65 auto antibodies
* Occurrence of type 1 diabetes in first degree relatives
* Anaemia
* Pregnancy and/or breast feeding
* Treatment with medication affecting insulin secretion
* non-compliance

Withdrawal criteria

* The subject may withdraw at will at any time
* Pregnancy discovered during the trial
* Severe illness
* Unacceptable side effects
* If self-measured fasting plasma glucose on three consecutive days exceeds 15 mM, the result is repeated in an immediately scheduled visit, and no treatable intercurrent cause for the hyperglycaemia can be found.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-02; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kasper Aaboe, MD, Principal Investigator — Gentofte University Hospital
Locations (1):
- Gentofte Hospital, Hellerup, Denmark

REFERENCES:
- [Derived] Aaboe K, Akram S, Deacon CF, Holst JJ, Madsbad S, Krarup T. Restoration of the insulinotropic effect of glucose-dependent insulinotropic polypeptide contributes to the antidiabetic effect of dipeptidyl peptidase-4 inhibitors. Diabetes Obes Metab. 2015 Jan;17(1):74-81. doi: 10.1111/dom.12395. Epub 2014 Oct 26. PMID 25243647

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from Jan. 2008 to Dec 2009 through out-patient clinic and advertisement
Groups:
- Placebo: Placebo treatment
Period: Overall Study
Arm/Group | Placebo | Januvia
Started | 24 | 25
Completed | 24 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Januvia | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 25 | 48
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 60 [31 to 72] | 60 [39 to 64] | 60 [31 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 13 | 13 | 26
Region of Enrollment [Number; unit: participants]
  Denmark | 24 | 25 | 49

OUTCOME MEASURES:

1. Primary Outcome: the Relative Increase in Meal-induced Total GLP-1 Secretion
Description: Patients will be followed for 12 weeks with three meal test examinations; before treatment, after 1 week of treatment and after 12 weeks of treatment. Primary outcome is AUC GLP-1 (pM x 120 as stated).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: pM x 120 min
Arm/Group | Placebo | Januvia
Number analyzed (Participants) | 12 | 12
pM x 120 min | 2591 (358) | 3959 (877)

2. Primary Outcome: Restoration of the Insulinotropic Effect of GIP
Description: Restoration of the insulinotropic effect of GIP measured as the relative increase in GIP induced amplification of the late phase insulin secretion (AUC) response to glucose. Patients will be followed for 12 weeks with examinations after 1 and after 12 weeks of treatment.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: pM x 120 min
Arm/Group | Placebo | Januvia
Number analyzed (Participants) | 12 | 13
pM x 120 min
  After 1 week | 17.8 (3.0) | 21.3 (4.3)
  After 12 weeks | 19.7 (3.7) | 30.0 (6.2)

3. Secondary Outcome: Examination of GLP-2, Somatostatin, Glucagon, Peptide-YY and Two Glycaemic Control Parameters (HbA1c and Fasting Plasma Glucose)
Description: Secondary objectives are examination of GLP-2, somatostatin, glucagon, peptide-YY and two glycaemic control parameters (HbA1c and fasting plasma glucose). Patients will be followed for 12 weeks with three examinations; before, during and after the treatment
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Placebo: No adverse events recorded
- Januvia: Active treatment. No adverse events recorded
Arm/Group | Placebo | Januvia
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less